CLINICAL TRIAL: NCT02872337
Title: One-on-One Physical Therapy Education Improves Postoperative Function and Patient Satisfaction After TJA
Brief Title: Pre-operative One-on-One Physical Therapy Education Improves Postoperative Function and Patient Satisfaction After Total Joint Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-306
Record Dates: First submitted 2016-08-01; First posted 2016-08-19 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Intervention): PreopPT Group (Experimental): This group will undergo the group preoperative education session. Following this session (intervention) this group underwent a one-time, one-on-one preoperative PT session. They also were given access to a web-based microsite which was customized to surgeon
  Interventions: Behavioral: Preoperative Physical Therapy Session; Behavioral: Group Preoperative Education Session (per the standard of care)
- Control (standard of care): No PreopPT Group (Placebo Comparator): This group underwent the current of standard of care at our institution. This only includes the group preoperative education session. No further preoperative education was given.
  Interventions: Behavioral: Group Preoperative Education Session (per the standard of care)

INTERVENTIONS:
Behavioral: Preoperative Physical Therapy Session — This was a one-on-one preoperative physical therapy session on preoperative education. These patients were also given access to a surgery specific web-based microsite
  Arms: Experimental (Intervention): PreopPT Group
Behavioral: Group Preoperative Education Session (per the standard of care)

SUMMARY:
The purpose of this study was to evaluate the efficacy of a one-time, preoperative physical therapy protocol on postoperative (1) discharge disposition, (2) pain, function and stiffness and (3) patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be required to meet the following inclusion criteria in order to participate:

  * Unilateral Primary Knee OA or Hip OA
  * Patients at least 18 years old up to 85.
  * Undergoing surgery with one of the following study surgeons
  * Able to independently ambulate ≥ half a block with or without assistive device
  * Able to independently perform non-reciprocal stairs with or without assistive device/rails
  * Patients that plan to D/C home post TKA / THA
  * Patients that speak English only.

Exclusion Criteria:

* Rheumatoid arthritis
* Psoriatic arthritis
* Juvenile rheumatoid arthritis
* Knee or Hip revisions
* Patients under 18 years of age
* Patients unwilling or unable to complete PRO instrument or study questionnaires at the specified study time points pre-operatively or post-operatively
* Bilateral TKA and THA
* Uni-condylar knee arthroplasty or Hip resurfacing
* Patellar reconstruction
* Patient on disability, workman's compensation
* Patients unwilling to participate in PEdPTWP and/or Patient education class and booklet.
* Patients that plan to D/C to rehabilitation center post TKA and THA
* Patients that do not speak English
* Patients that do not have access to computer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of In-patient Physical Therapy visits required to meet hospital discharge criteria PT | Through Study Completion, an average of 3 days
  This included a review of the hospital database for hospital discharge time. At this institution PT discharge is defined as the ability to (1) independently transfer, (2) independently ambulate approximately 150 feet and (3) independently negotiate stairs (4) independent with home exercise program and activities of daily living.
  All of this data was recorded from hospital records

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | This standard patient reported outcome was filled out preoperatively or at six weeks postoperatively
  This standard patient reported outcome was filled out preoperatively or at six weeks postoperatively
Patient Satisfaction Scores | from two weeks prior to surgery until 6 weeks after surgery
  Patient satisfaction was measured by a series of patient administered questionnaires at various stages of the study. All satisfaction questions, with the exception of the utilization of the microsites [Yes/No], were asked via a visual analogue scale to disagree or agree with given statements [0-5, where 0 was strongly disagree, 3 was neutral and 5 was strongly agree]. Patients unable to complete any forms at the time of the appointment completed the form over the phone with a co-investigator.
Time to meet Physical Therapy discharge criteria | Time from Surgery to meeting PT discharge criteria, an average of 3 days
  At this institution PT discharge is defined as the ability to (1) independently transfer, (2) independently ambulate approximately 150 feet and (3) independently negotiate stairs (4) independent with home exercise program and activities of daily living.
Hospital Length of Stay | Time from Surgery until Hospital Discharge, an average of 2-3 days
  collected from a hospital database